CLINICAL TRIAL: NCT05211817
Title: Physical Activity and Nutrition Program in the Prevention and Treatment of Obesity, Mechanisms of Obesity and Its Comorbidities
Brief Title: Research on Prevention, Intervention and Mechanisms of Obesity and Its Comorbidities
Acronym: Obesity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Slovak Academy of Sciences (Other Government)
Collaborators: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Barbara Ukropcová, MD, PhD, Professor, Slovak Academy of Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 313011V344
Record Dates: First submitted 2021-11-02; First posted 2022-01-27 (Actual); Last update posted 2022-01-27 (Actual); Status verified 2022-01

CONDITIONS: Obesity; Exercise; Nutrition, Healthy
MeSH Terms: conditions — Obesity; Motor Activity | interventions — Carnosine

STUDY DESIGN:
Intervention Model Description: Randomised controlled trial with complex lifestyle intervention and carnosine supplementation.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Block randomisation for carnosine, identically looking control and intervention treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Complex Intervention with Carnosine (Experimental): Obese middle aged individuals will be subjected to 3 month complex lifestyle intervention including exercise (3 times per week) nutritional (weekly consultation) and psychological (monthly) interventions combined with oral administration of carnosine in dose 2g per day.
  Interventions: Behavioral: Complex lifestyle intervention; Dietary Supplement: Carnosine
- Complex Intervention with placebo (Experimental): Obese middle aged individuals will be subjected to 3 month complex lifestyle intervention including exercise (3 times per week) nutritional (weekly consultation) and psychological (monthly) interventions combined with oral administration of identically looking placebo.
  Interventions: Behavioral: Complex lifestyle intervention
- Without complex intervention with carnosine (Experimental): Obese middle aged individuals will be subjected to standard clinical procedure without lifestyle interventions. Oral administration of carnosine in dose 2g per day will be provided.
  Interventions: Dietary Supplement: Carnosine
- Without complex intervention with placebo (No Intervention): Obese middle aged individuals will be subjected to standard clinical procedure without lifestyle interventions. Oral administration of identically looking placebo will be provided.

INTERVENTIONS:
Behavioral: Complex lifestyle intervention — Volunteers will undergo a 3-month comprehensive lifestyle modification, consisting of a combined aerobic-strength training intervention, nutritional and psychological counseling. Regular examinations (body weight, waist circumference, body composition by bioimpedance) will be performed every week. Probands in the intervention and control groups will have the opportunity to participate in a long-term program of physical activity at BMC SAS after the end of the study.
  Arms: Complex Intervention with Carnosine; Complex Intervention with placebo
Dietary Supplement: Carnosine — 3 months carnosine supplementation (2 g per day) will be given in parallel with a complex lifestyle modification. Carnosine is a dipeptide of beta-alanyl l-histidine, which is found in skeletal muscle and in certain areas of the brain. It is a well-tolerated and approved food supplement in Slovakia. Scientists have extensive experience with the administration of carnosine (deCourten, Ukropcová et al, Obesity 2015 https://doi.org/10.1002/oby.21434; Schon, Ukropcova et al, 2019 DOI: 10.3390 / nu11061196 and others). Carnosine has the potential to positively affect glucose metabolism, and improve the adaptive response to exercise training interventions.
  Arms: Complex Intervention with Carnosine; Without complex intervention with carnosine

SUMMARY:
Obesity and lack of physical activity are associated with an increased risk of many chronic diseases and accelerate the processes associated with aging. Weight reduction and physical fitness are health benefits of long-term and comprehensive lifestyle modification based on nutritional habits, increased physical activity and psychotherapy. A healthy lifestyle is the basis for the prevention and treatment of obesity. However, conditions for the prescription of physical activity, nutrition and psychotherapy have not been established in our healthcare system. The aim of the project is to determine the effects of a 3-month complex intervention with/without carnosine (including aerobic/strength training, nutritional and psychological counseling) on body composition, physical fitness and circulating biochemical characteristics. Molecular biomarkers can be a very useful diagnostic markers as well as a parameter for monitoring the effectiveness of a complex lifestyle intervention. Long-term follow-up and inclusion in long-term programs will be offered to all study probands who are interested.

DETAILED DESCRIPTION:
Training is combining one 60min session of aerobic training with two 1-hour weekly lessons of aerobic strength training composed of 25 minutes, 60-70% 1RM, training the large muscle groups and 25 minutes of rowing or stationary biking. Starting with warm-up and stretching cool down at the end. The individualized training program will be based on the actual patients physical fitness (VO2max, bicycle spiroergometry) and muscle strength (dynamometry). The training will take place in small groups of 4-5 volunteers. There will be 15-minute breaks for ventilation and surface disinfection between training sessions. All coaches of the Center are vaccinated. The aim is to provide a safe environment for training, in order to increase physical fitness and reduce the weight of obese patients. The center has experience with full-time and online trainings (via the publicly available Facebook BMC SAS as well as through the ZOOM platform) http://www.biomedcentrum.sav.sk/centrum-pohybovej-aktivity/

The nutritional intervention will be carried out by nutrition specialists with the use of individual and group counseling, which enables the individualized dietary prescription. Coaching will take place in person in groups of 5-10 probands (BMC SAS, with a frequency of once a month, in accordance with the current epidemiological situation), resp. by phone / online, with a frequency of once a week.

Psychological counseling will be provided by clinical psychologists. Individual and group form, with a frequency of at least once per month. Psychological counseling will focus on identifying the triggers of inappropriate eating behavior and influencing them, as well as supporting the development of new, healthier habits.

3 months carnosine supplementation (2 g per day) will be provided as described elsewhere.

ELIGIBILITY:
Inclusion Criteria:

* sedentary men and women (approximately 1:1) aged 25-45 years, BMI 28-38 kg/m2
* absence of chronic diseases and regular pharmacotherapy intake
* capable to complete a training intervention (assessment by a cardiologist)
* signed informed consent
* absence of any psychological, sociological or geographical factors that could jeopardize participation in the study
* Vaccination against SARS-CoV-2 with one of the approved vaccines available in Slovakia (at least 2 weeks after the last dose) and regular PCR testing during the study.

Exclusion Criteria:

* any chronic disease (oncological, cardiovascular, neurological, liver, kidney or other diseases and its acute complications at the discretion of the doctor);
* No cooperation of probands;
* insufficient functional capacity - the presence comorbidities or disorders of the musculoskeletal system, which makes it impossible to complete the training program (assessment by cardiologist, or orthopedist or other specialist);
* smoking, alcohol or drugs abuse;
* non-compliance with epidemiological measures;
* absence of complete vaccination with SARS-CoV-2 vaccine;
* presence of a pacemaker or metal implants (contraindication for magnetic resonance imaging).

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Intervention induced change in abdominal adiposity | 3 months
  Body fat composition will be measured by bioelectrical impedance analysis and presented in percentage.
Intervention induced change in VO2max. | 3 months
  Maximal aerobic capacity will be measured by testing physical performance on a bicycle ergometer. Results will be presented as mL/(kg·min) units.
Intervention induced change in abdominal muscle mass | 3 months
  Changes in the abdominal muscle mass will be measured by Magnetic resonance imaging (MRI).
Intervention induced change in muscle strength. | 3 months
  Muscle strength will be measured by handheld dynamometer.
Intervention induced change in glucose level and glucose metabolism. | 3 months
  Fasting glucose level measurement and glucose tolerance test will be provided for volunteers.
Intervention induces change in lipid profile. | 3 months
  Measurement of total cholesterol, HDL, LDL, VLDL and triglycerides will be performed from the blood samples.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Ukropcova, Prof., Principal Investigator — Biomedical Research Centre SAS
Locations (1):
- Biomedical Research Center Slovak Academy of Sciences, Bratislava, Slovakia

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, CSR
Time Frame: 31.12.2025 indefinitely
Access Criteria: In principle to all researchers working in the area. Requests will be reviewed by Prof. Barbara Ukropcova.